CLINICAL TRIAL: NCT02400463
Title: Pilot Study of Ruxolitinib in Secondary Hemophagocytic Syndrome
Brief Title: A Pilot Study of Ruxolitinib in Secondary Hemophagocytic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.112; HUM00092921 (Other: University of Michigan)
Record Dates: First submitted 2015-01-22; First posted 2015-03-27 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Hemophagocytic Syndrome (HPS)
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib 15 mg by mouth twice daily.
  For patients unable to ingest tablets, ruxolitinib suspended in water may be administered through a nasogastric (NG) or percutaneous endoscopy gastrostomy (PEG) tube.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib

SUMMARY:
This is a pilot study to determine the efficacy of Ruxolitinib in secondary hemophagocytic syndrome. The primary objective is to assess the efficacy of ruxolitinib 15 mg PO twice daily in patients with HPS. The primary endpoint is overall survival at two months.

DETAILED DESCRIPTION:
Hemophagocytic Syndrome (HPS) is a disorder characterized by pathological activation of the immune system resulting in a systemic disorder characterized by excessive cytokine production and macrophage activation, culminating in cytopenias and evidence of hemophagocytosis on tissue specimens. The disorder can be sporadic or familial due to one of several mutations and is primarily seen in the pediatric population, with a reported incidence of 1 case per 3000 admissions. The actual incidence in adults is unknown and can be rarely sporadic, or secondary to viral infections, malignancy, or autoimmune disease.

HPS is a universally fatal disease if untreated. In adults, the median survival has been reported to be less than 2 months if diagnosis and treatment is delayed. Adult patients are treated with pediatric protocols with early institution of etoposide and steroids and consolidation with allogeneic stem cell transplant in appropriately selected patients if a familial form is identified. Other treatment strategies have been attempted, including rituximab, infliximab, entaracept, tocilizumab, and alemtuzumab. These anecdotal reports highlight the therapeutic potential of cytokine-targeted therapies in this disorder.

This is a pilot study to determine the efficacy of Ruxolitinib in secondary hemophagocytic syndrome. The primary objective is to assess the efficacy of ruxolitinib 15 mg PO twice daily in patients with HPS. The primary endpoint is overall survival at two months.

Patients will receive Ruxolitinib at 15 mg twice daily orally either on an empty stomach or with food for 4 weeks (28 days) in a 4 week (28 day) cycle. Ruxolitinib will be administered in continuous 28-day cycles.

In the absence of treatment delays or cessation due to adverse events, treatment may continue indefinitely or until one of the following criteria applies:

* Disease progression.
* Intercurrent illness that prevents further administration of treatment.
* The investigator considers it, for safety reasons, to be in the best interest of the patient.
* Unacceptable adverse events such as any toxicity or other issue that causes a delay of study drug administration by more than 4 weeks.
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.
* Patient decision to withdraw from treatment (partial consent) or from the study (full consent.
* Death.

Patients will be followed for toxicity for 30 days after treatment has been discontinued or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients, or their legally authorized representative, must voluntarily provide written IRB-approved informed consent.
* Males and females, 18 years of age or older at the time of enrollment.
* Patients must meet the diagnostic criteria for HPS (at least 5 of the following): fever, splenomegaly, cytopenia involving ≥2 cell lines (Hemoglobin <9 g/dL; platelets <100,000/μL; absolute neutrophil count <1000/μL), hypertriglyceridemia or hypofibrinogenemia, tissue demonstration of hemophagocytosis, low or absent NK (Natural Killer) cell activity, serum ferritin ≥3000 ug/L, soluble IL-2 receptor (CD25) >2400 U/mL.
* In the investigator's opinion, the patient has the ability to participate fully in the study, and comply with all its requirements.

Exclusion Criteria:

* CNS (Central Nervous System) involvement
* Malabsorption
* Known secondary HPS (Hemophagocytic Syndrome) that is otherwise treatable (e.g. non-Hodgkin's lymphoma).
* Pregnant or lactating female: all females of child-bearing potential must have a negative serum pregnancy test within 7 days of treatment; lactating females must discontinue breast feeding.
* Estimated creatinine clearance <15mL/min
* Has received any prior systemic therapy, excluding corticosteroids, within 7 days (or 5 half-lives) of treatment.
* No active malignancy at the time of enrollment, except nonmelanoma skin cancers or carcinoma in situ. Patients with a prior history of malignancy are eligible if their malignancy has been definitely treated or is in remission and does not require ongoing adjuvant or cancer-directed therapies.
* Active hepatitis B or hepatitis C or known HIV infection
* Known (and biopsy-confirmed) liver cirrhosis; or, a reported history of liver cirrhosis with a Model for End-stage Liver Disease (MELD) score >20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, M.D., Principal Investigator — Int Med-Hematology/Oncology - Faculty and Staff
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Ahmed A, Merrill SA, Alsawah F, Bockenstedt P, Campagnaro E, Devata S, Gitlin SD, Kaminski M, Cusick A, Phillips T, Sood S, Talpaz M, Quiery A, Boonstra PS, Wilcox RA. Ruxolitinib in adult patients with secondary haemophagocytic lymphohistiocytosis: an open-label, single-centre, pilot trial. Lancet Haematol. 2019 Dec;6(12):e630-e637. doi: 10.1016/S2352-3026(19)30156-5. Epub 2019 Sep 16. PMID 31537486
- See also: The Lancet Haematology, VOLUME 6, ISSUE 12, E630-E637, DECEMBER 01, 2019 — https://doi.org/10.1016/S2352-3026(19)30156-5

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 38 [29 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 2 Months
Description: Number of Patients Alive at 2 Months after the first administration of ruxolitinib.
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Percentage of Patients With a Response to Treatment With Ruxolitinib
Description: Complete response is defined as complete normalization of all quantifiable symptoms and laboratory abnormalities. A partial response is defined as at least a 25% improvement in two or more quantifiable symptoms/laboratory markers.
Time Frame: 2 Months
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 6
percentage of participants | 100

3. Secondary Outcome: Duration of Response
Description: Duration will be calculated from the date of the determination of partial response or better until the date of progression, death, or additional non-protocol therapy.
Time Frame: Up to 3 years (Due to funding and other constraints, participant follow-up was discontinued in 2020. Thus, not all participants were followed for a full three years.)
Measure: Median (Full Range); unit: months
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 6
months | 17.25 [3.5 to 35.5]

4. Secondary Outcome: Progression Free Survival Time
Description: Progressive Disease is defined as at least a 50% worsening in two or more quantifiable laboratory markers. Calculated from the first administration of ruxolitinib until the date of progression or death.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 6
months | 17.25 [3.5 to 35.5]

5. Secondary Outcome: Regimen Related Toxicities
Description: Incidence and grade of adverse events (AEs) unlikely, possibly or probably related to treatment (tx) with ruxolitinib. Graded per Common Terminology Criteria for Adverse Events (CTCAE) v.4. Grade refers to the severity of the AE, from mild (grade 1) to life-threatening (grade 4).
Time Frame: Up to 30 days after last treatment administration
Measure: Number; unit: Adverse Events
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 6
Adverse Events
  Grade 1 | 5
  Grade 2 | 3
  Grade 3 | 1
  Grade 4 | 1

ADVERSE EVENTS:
Time Frame: Up to 30 days after last treatment administration (13.5 months)
Arm/Group | Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=6)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (4)
Localized edema (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (3)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02400463/Prot_SAP_000.pdf